CLINICAL TRIAL: NCT02930395
Title: Blood Biomarkers for the Management of Concussion in Professional Rugby Players
Acronym: RUGBYPROS100B
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: World Rugby Research Unit (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-0282; DC-2016-2742 (Other: DC-2016-2742)
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Concussion; Professional TOP14 Rugby Players
Keywords: Concussion; Professional rugby players; S100B
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- professional rugby players
  Interventions: Procedure: serum S100B assay

INTERVENTIONS:
Procedure: serum S100B assay

SUMMARY:
In the past 20 years, the incidence of concussion in direct contact sports has significantly increased. The incidence of concussion in rugby players ranges between 8 to 17 episodes / 1000 playing hours. A recent study published by the French Rugby Federation (FFR) and the National Rugby League (LNR) showed similar results. The latter study was performed analyzing the French "TOP14", which includes 14 teams participating in professional rugby championships. At least two concussions were diagnosed each week. Despite the recent evidence, cognitive assessment remains the only means to determine whether or not players experiencing concussions can return to the game or not.

DETAILED DESCRIPTION:
The possible evolution of neuro-vascular damage and its biological consequences are currently overlooked. The Head Injury Assessment (HIA) is the current gold standard used by the national Rugby Medical Authorities in accordance with international safety protocols. The HIA protocol relies on neurological or neuropsychological endpoints, potentially subjective or not ensuring sufficient sensitivity. As a result, defining the immediate and long-term pathophysiological consequences of concussions remains challenging. The introduction of an objective blood test to detect the presence and the evolution overtime of neuro-vascular damage could represent a pairing approach filling a sensitive gap in the management of concussed players. Recent evidence has proposed the use of serum biomarkers aiding post-concussion management . Remarkably, serum biomarkers of neuro-vascular functions are currently being used in emergency room settings. Serum levels of the brain protein S100β were demonstrated to have an excellent negative predictive value for neurovascular damage after mild traumatic brain injury (mTBI). Measurement of blood S100β was proposed as a tool to grade TBI, limiting unnecessary CT scan examinations in emergency cases . However, whether the use of serum makers of neuro-vascular damage could benefit the management of sport-related concussion remains unclear. Moreover, repeated concussions have been linked to an increased risk of Alzheimer's disease, Multiple Sclerosis and Parkinson's disease . Serum biomarkers could be of diagnostic and prognostic value, facilitating return to play decisions or predicting lingering risks of cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Players age > 18 years old.
* Players routinely managed by the medical staff of collaborative rugby teams. Availability of clinical data, age, body mass index, brain performance, previous HIA scores, history of concussions.
* Players must agree with all of the aspects of the research. Players must consent for a baseline blood draw before the season starts and follow up sampling after concussions

Exclusion Criteria:

* Adverse players' life style (e.g., alcohol consumption, medications or chronic drug regimens) or pathological conditions associated with abnormal S100β levels (e.g., S100 genetic variants, cutaneous infections, brain tumor, auto-immune disorders, or hyper-lymphocytosis).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Professional rugby players
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
significance of S100β/HIA score in the early management of concussion | at day 1
significance of unveiling novel markers of long-term brain cell damage in rugby players | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Vincent SAPIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- See also: Utility of S100B Serum Level for the Determination of Concussion in Male Rugby Players — http://www.ncbi.nlm.nih.gov/pubmed/27430504
- See also: Systematic review of clinical studies examining biomarkers of brain injury in athletes after sports-related concussion — http://www.ncbi.nlm.nih.gov/pubmed/25254425